CLINICAL TRIAL: NCT02220491
Title: A Randomized Phase II Study of 20 Gy in 5 Fractions Whole Brain Radiotherapy Versus 15 Gy in 1 Fraction Volumetric Modulated Arc Therapy for One to Ten Brain Metastases
Brief Title: Whole Brain Radiotherapy Versus Volumetric Modulated Arc Therapy for Brain Metastases
Acronym: Amadeus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H14-02032
Record Dates: First submitted 2014-08-15; First posted 2014-08-20 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole-brain radiotherapy (Active Comparator): All subjects will have a non-contrast CT scan using a slice thickness of 2.5mm or less.
  The Brain contour will be generated using the segmentation wizard and edits as required.
  PTV_Brain is an expansion of the Brain by 5mm. 99% of PTV_Brain is to be covered by 95% of 20 Gy in 5 fractions using 6-10 MV photons in a parallel-opposed pair lateral beam arrangement.
  Interventions: Radiation: Whole-brain radiotherapy
- Single-fraction radiotherapy (Experimental): Immobilized in the mask, the subject will be imaged for radiotherapy planning with a CT slice thickness of 1.25 mm or less and an axial resolution of < 0.7 mm (CT field of view < 35 cm). Subjects that require contrast with GFR 45-59 will have pre-hydration, contrast dose modification and/or Mucomyst administration to preserve renal function, according to standard practice for radiological imaging at the institution.
  Interventions: Radiation: Single-fraction radiotherapy

INTERVENTIONS:
Radiation: Single-fraction radiotherapy — Volumetric modulated arc therapy (VMAT) delivering 15 Gy in one fraction to brain metastases
  Arms: Single-fraction radiotherapy
Radiation: Whole-brain radiotherapy — Whole brain radiotherapy delivering 20 Gy in five fractions to brain metastases
  Arms: Whole-brain radiotherapy

SUMMARY:
Patients with brain metastases with expected life expectancy of 3-6 months are typically treated with radiotherapy to the whole brain giving a dose of 20 Gy over a 5 day period. This study will compare this with volumetric modulated arc therapy (VMAT) which is capable of delivering 15 Gy in one single session to identified disease within the brain but sparing the normal surrounding brain tissue. Primarily the study will assess whether it is possible to recruit sufficient patient numbers to a trial of this type. It will also compare effectiveness, side effects and quality of life between the two treatment methods.

DETAILED DESCRIPTION:
This is a Phase II prospective clinical trial. Pre treatment evaluations include estimation of life expectancy, Creatinine (GFR) and MRI brain with contrast. An assessment of cognitive function using Montreal Cognitive Assessment questionnaire, assessment of daily living activities using the Modified Barthel's index and quality of life assessment using EORTC QLQ-PAL-15 & BN-20 questionnaires will be performed in clinic. Karnofsky Performance Status will also be assessed by the clinician. If all assessments are within the eligibility criteria then the patient can be recruited. Before treatment begins a history documenting baseline symptoms using NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 and a neurological examination documenting baseline deficits must be obtained.

If patient is randomized to standard treatment of whole brain radiotherapy (WBRT) then subjects will have a non-contrast CT scan using a slice thickness of 2.5 mm or less to plan radiotherapy. If patient are randomized to single fraction radiotherapy then a contrast CT will be used as this aids in identifying metastatic tumours within the brain. Also for the single fraction arm if a contrast-enhanced diagnostic MRI was obtained ≤ 10 days before the CT planning scan, with a single-plane high-resolution sequence or low-resolution sequences in two planes, it can be used for treatment planning. If the contrast-enhanced diagnostic MRI was obtained > 10 days before the CT planning scan or there is no diagnostic MRI, the subject requires a gadolinium-enhanced, high-resolution MRI sequence for fusion in the treatment planning system. During treatment, patients will have daily online cone beam CT scans to apply setup corrections to ensure treatment accuracy. To ensure minimal movement during radiotherapy all subjects will be immobilized lying on their back in a plastic headshell with an integrated bite block.

For subjects in the single-fraction arm that are not requiring steroids before radiotherapy, dexamethasone 8 mg 1 hour before the radiotherapy and for 5 days afterwards is required. For subjects in the single-fraction arm that are requiring corticosteroids for symptom management before radiotherapy, dexamethasone 8 mg before treatment and 8 mg 2 times daily for 2 days is required. Beginning three days after radiotherapy, a taper back to the pre-radiotherapy dose can be done swiftly over 4-6 days. However, for subjects who have been on dexamethasone for more than 2 weeks at this time point, slow tapering from the pre-radiotherapy dose using decrements of 0.5 - 2 mg every 3-5 days should be used to prevent a hypocortisolemia. For subjects in the 5-fraction arm, corticosteroids will be prescribed according to the preference of the treating radiation oncologist. Anti-sickness medication and steroids will be prescribed are required before each fraction in both arms.

Following therapy completion, all patients will be seen at 6 weeks, 3, 6, 9 and 12 months. At each visit history and neurological examination will be performed. Cognitive Function, Karnofsky Performance Status, Quality of life and Adverse Events will all be assessed and recorded. Activities of Daily Living and steroid use will be assessed by telephone consultation every 4 weeks (monthly) for 1 year. Steroid use will be confirmed by evaluating the pharmacy prescription database.

Patients will have contrast-enhanced MRI brain at every time point with a creatinine 1 week before each MRI to ensure safety of intravenous contrast administration. Steroid use will be recorded in a patient diary for first 6 weeks post treatment and monthly by telephone discussion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Pathologically confirmed solid malignancy
* 1-10 brain or brainstem metastases on MRI with a maximum of 4 cm diameter
* Documented extracranial disease
* Anticipated median survival 3-6 months (Graded Prognostic Assessment: Appendix I)
* Available for regular clinical and imaging follow up (< 1 hour from a cancer centre)
* Montreal Cognitive Assessment score ≥ 20 (Appendix II)
* Karnofsky Performance Score (KPS) ≥ 70 (Appendix III)
* Barthel Activities of Daily Living score ≥ 90 (Appendix IV)
* Able to complete EORTC quality of life questionnaires (Appendix V)

Exclusion Criteria:

* A metastasis located within 5 mm of the optic nerves or optic chiasm
* Requiring craniotomy to relieve mass effect
* Cytotoxic systemic therapy administered within one week before radiotherapy or planned within one week after radiotherapy
* Neurological decline since starting corticosteroids
* Metastatic germinoma, small cell carcinoma, multiple myeloma, lymphoma or leukaemia
* Systemic lupus erythematosis, scleroderma, or other connective tissue disorders not in remission
* Multiple sclerosis
* Glomerular Filtration Rate < 45 ml/minute
* Contra-indications to MRI
* Pregnancy
* AST, ALT or Bilirubin > 3 times upper limit of normal
* Haemorrhagic Metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Accrual | 8 months
  The time of accrual of 20 subjects will be recorded in months from the official study opening at each cancer centre until the 20th patient is accrued. The rate of accrual will be calculated by dividing the number of patients by the number of months it took to accrue them

SECONDARY OUTCOMES:
Intracranial disease control | 3 months
  All subjects who complete radiotherapy and have imaging at 6 weeks will be considered evaluable for response. Those who exhibit objective disease progression on imaging before 6 weeks will also be considered evaluable for response.

OTHER OUTCOMES:
Compare the use of corticosteroids | Every 4 weeks for 1 year
  The subjects' use of corticosteroids will be recorded in a diary for the first 6 weeks and assessed monthly with phone follow-up. The amount and pattern of corticosteroid use will be compared between the two arms of the study.
Compare the incidence of retreatment with cranial radiotherapy | 3 months
  Subjects with new brain metastases can be treated in a number of ways if their performance status remains good. If 3 months have passed since their initial treatment and there are 1-10 new metastases, subjects can receive the study treatment with 15 Gy in 1 fraction again. However, if the new brain metastases are detected within 3 months or there are more than 10 new brain metastases, subjects must have WBRT, rather than treatment to the metastases alone. Subjects with progression or relapse of a treated brain metastasis can be considered for surgery, retreatment with radiosurgery or retreatment with WBRT. Subjects with poor performance status should be considered for best supportive care.
Compare the incidence of acute and late side effects | 6 weeks, 3 months, 6 months, 9 months, 12 months
  The study will use the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) for grading of acute and late side effects. The incidence of the various side effects will be compared between the two arms.
Compare the time to decline in activities of daily living using the Modified Barthel Index | Every 4 weeks for 1 year
  The Modified Barthel index will be administered at baseline and at each follow-up visit. The scores will be recorded and analysed. The minimum clinically important difference for this scale is 10 points.
Compare the time to decline in Karnofsky Performance Status < 70 | 6 weeks, 3 months, 6 months, 9 months, 12 months
  The KPS will be recorded at each clinic visit. The patient will be regarded as having had a decline in KPS when it falls below 70, at which time subjects are no longer independent.
Compare the time to decline in cognition | 6 weeks, 3 months, 6 months, 9 months, 12 months
  The MoCA questionnaire will be administered at baseline and at each follow-up visit (Appendix II). The score will be recorded and analysed. A decline in MOCA score of 3 is considered to be clinically significant.
Time to decline in quality of life | 6 weeks, 3 months, 6 months, 9 months, 12 months
  The EORTC QLQ-PAL-15 will be administered at baseline and at each follow-up visit. The EORTC BN-20 (brain-specific) quality of life questionnaire will be administered at baseline and at each follow-up visit. The quality of life questionnaire scores will be recorded and analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Nichol Alan, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Mekhail T, Sombeck M, Sollaccio R. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. Curr Oncol Rep. 2011 Aug;13(4):255-8. doi: 10.1007/s11912-011-0180-1. No abstract available. PMID 21584645
- [Background] Soon YY, Tham IW, Lim KH, Koh WY, Lu JJ. Surgery or radiosurgery plus whole brain radiotherapy versus surgery or radiosurgery alone for brain metastases. Cochrane Database Syst Rev. 2014 Mar 1;2014(3):CD009454. doi: 10.1002/14651858.CD009454.pub2. PMID 24585087
- [Background] Soffietti R, Kocher M, Abacioglu UM, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Mueller RP, Tridello G, Collette L, Bottomley A. A European Organisation for Research and Treatment of Cancer phase III trial of adjuvant whole-brain radiotherapy versus observation in patients with one to three brain metastases from solid tumors after surgical resection or radiosurgery: quality-of-life results. J Clin Oncol. 2013 Jan 1;31(1):65-72. doi: 10.1200/JCO.2011.41.0639. Epub 2012 Dec 3. PMID 23213105
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Rodrigues G, Warner A, Zindler J, Slotman B, Lagerwaard F. A clinical nomogram and recursive partitioning analysis to determine the risk of regional failure after radiosurgery alone for brain metastases. Radiother Oncol. 2014 Apr;111(1):52-8. doi: 10.1016/j.radonc.2013.11.015. Epub 2014 Jan 17. PMID 24444529
- [Background] Tsao MN, Lloyd N, Wong RK, Chow E, Rakovitch E, Laperriere N, Xu W, Sahgal A. Whole brain radiotherapy for the treatment of newly diagnosed multiple brain metastases. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD003869. doi: 10.1002/14651858.CD003869.pub3. PMID 22513917
- [Background] Andrews DW, Scott CB, Sperduto PW, Flanders AE, Gaspar LE, Schell MC, Werner-Wasik M, Demas W, Ryu J, Bahary JP, Souhami L, Rotman M, Mehta MP, Curran WJ Jr. Whole brain radiation therapy with or without stereotactic radiosurgery boost for patients with one to three brain metastases: phase III results of the RTOG 9508 randomised trial. Lancet. 2004 May 22;363(9422):1665-72. doi: 10.1016/S0140-6736(04)16250-8. PMID 15158627
- [Background] Shaw E, Scott C, Souhami L, Dinapoli R, Bahary JP, Kline R, Wharam M, Schultz C, Davey P, Loeffler J, Del Rowe J, Marks L, Fisher B, Shin K. Radiosurgery for the treatment of previously irradiated recurrent primary brain tumors and brain metastases: initial report of radiation therapy oncology group protocol (90-05). Int J Radiat Oncol Biol Phys. 1996 Feb 1;34(3):647-54. doi: 10.1016/0360-3016(95)02106-x. PMID 8621289
- [Background] Yamamoto M, Serizawa T, Shuto T, Akabane A, Higuchi Y, Kawagishi J, Yamanaka K, Sato Y, Jokura H, Yomo S, Nagano O, Kenai H, Moriki A, Suzuki S, Kida Y, Iwai Y, Hayashi M, Onishi H, Gondo M, Sato M, Akimitsu T, Kubo K, Kikuchi Y, Shibasaki T, Goto T, Takanashi M, Mori Y, Takakura K, Saeki N, Kunieda E, Aoyama H, Momoshima S, Tsuchiya K. Stereotactic radiosurgery for patients with multiple brain metastases (JLGK0901): a multi-institutional prospective observational study. Lancet Oncol. 2014 Apr;15(4):387-95. doi: 10.1016/S1470-2045(14)70061-0. Epub 2014 Mar 10. PMID 24621620
- [Background] Clark GM, Popple RA, Young PE, Fiveash JB. Feasibility of single-isocenter volumetric modulated arc radiosurgery for treatment of multiple brain metastases. Int J Radiat Oncol Biol Phys. 2010 Jan 1;76(1):296-302. doi: 10.1016/j.ijrobp.2009.05.029. PMID 19836151
- [Background] Stieler F, Fleckenstein J, Simeonova A, Wenz F, Lohr F. Intensity modulated radiosurgery of brain metastases with flattening filter-free beams. Radiother Oncol. 2013 Dec;109(3):448-51. doi: 10.1016/j.radonc.2013.10.017. Epub 2013 Nov 11. PMID 24231243
- [Background] Audet C, Poffenbarger BA, Chang P, Jackson PS, Lundahl RE, Ryu SI, Ray GR. Evaluation of volumetric modulated arc therapy for cranial radiosurgery using multiple noncoplanar arcs. Med Phys. 2011 Nov;38(11):5863-72. doi: 10.1118/1.3641874. PMID 22047350
- [Background] Karnofsky DA, Burchenal JH. The clinical evaluation of chemotherapeutic agents in cancer. In: MacLeod CM, editor. Evaluation of Chemotherapeutic Agents. Columbia University Press; 1949. p. 196.
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Background] Taphoorn MJ, Claassens L, Aaronson NK, Coens C, Mauer M, Osoba D, Stupp R, Mirimanoff RO, van den Bent MJ, Bottomley A; EORTC Quality of Life Group, and Brain Cancer, NCIC and Radiotherapy Groups. An international validation study of the EORTC brain cancer module (EORTC QLQ-BN20) for assessing health-related quality of life and symptoms in brain cancer patients. Eur J Cancer. 2010 Apr;46(6):1033-40. doi: 10.1016/j.ejca.2010.01.012. Epub 2010 Feb 22. PMID 20181476
- [Background] Caissie A, Nguyen J, Chen E, Zhang L, Sahgal A, Clemons M, Kerba M, Arnalot PF, Danjoux C, Tsao M, Barnes E, Holden L, Danielson B, Chow E. Quality of life in patients with brain metastases using the EORTC QLQ-BN20+2 and QLQ-C15-PAL. Int J Radiat Oncol Biol Phys. 2012 Jul 15;83(4):1238-45. doi: 10.1016/j.ijrobp.2011.09.025. Epub 2011 Dec 13. PMID 22172909
- [Background] Groenvold M, Petersen MA, Aaronson NK, Arraras JI, Blazeby JM, Bottomley A, Fayers PM, de Graeff A, Hammerlid E, Kaasa S, Sprangers MA, Bjorner JB; EORTC Quality of Life Group. The development of the EORTC QLQ-C15-PAL: a shortened questionnaire for cancer patients in palliative care. Eur J Cancer. 2006 Jan;42(1):55-64. doi: 10.1016/j.ejca.2005.06.022. Epub 2005 Sep 12. PMID 16162404
- [Background] Hsieh YW, Wang CH, Wu SC, Chen PC, Sheu CF, Hsieh CL. Establishing the minimal clinically important difference of the Barthel Index in stroke patients. Neurorehabil Neural Repair. 2007 May-Jun;21(3):233-8. doi: 10.1177/1545968306294729. Epub 2007 Mar 9. PMID 17351082
- [Background] Sperduto PW, Chao ST, Sneed PK, Luo X, Suh J, Roberge D, Bhatt A, Jensen AW, Brown PD, Shih H, Kirkpatrick J, Schwer A, Gaspar LE, Fiveash JB, Chiang V, Knisely J, Sperduto CM, Mehta M. Diagnosis-specific prognostic factors, indexes, and treatment outcomes for patients with newly diagnosed brain metastases: a multi-institutional analysis of 4,259 patients. Int J Radiat Oncol Biol Phys. 2010 Jul 1;77(3):655-61. doi: 10.1016/j.ijrobp.2009.08.025. Epub 2009 Nov 26. PMID 19942357
- [Derived] Raman S, Mou B, Hsu F, Valev B, Cheung A, Vallieres I, Ma R, McKenzie M, Beaton L, Rackley T, Gondara L, Nichol A. Whole Brain Radiotherapy Versus Stereotactic Radiosurgery in Poor-Prognosis Patients with One to 10 Brain Metastases: A Randomised Feasibility Study. Clin Oncol (R Coll Radiol). 2020 Jul;32(7):442-451. doi: 10.1016/j.clon.2020.02.001. Epub 2020 Feb 19. PMID 32085923